CLINICAL TRIAL: NCT07187024
Title: Efficacy of an Evidence-based Telehealth Intervention in Modifying Health Behaviors Associated With Post-Traumatic Osteoarthritis
Brief Title: Efficacy of an Evidence-based Telehealth Intervention in Modifying Health Behavior
Acronym: MIRROR_14
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Collaborators: University of North Carolina, Chapel Hill (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kenneth Cameron, Director of Orthopaedic and Sports Medicine Research, Keller Army Community Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RHC-A-19-034; 19KACH009 (Other: Keller)
Record Dates: First submitted 2020-07-07; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Post-traumatic Osteoarthritis; Knee Sprain; Knee Injuries
Keywords: Telehealth; Behavioral Intervention; PTOA
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The participants randomized to the intervention arm will be assigned to the mCare PTOA application, which consists of five modules that include basic information on joint health following injury, self-management strategies, weight management strategies, physical activity recommendations, and occupational management strategies to optimize joint health. These modules are delivered through the mCARE platform to a secure application on the participant's mobile device, provide interactive educational content on PTOA risk factors and strategies to mitigate those factors.
  Interventions: Behavioral: mCare PTOA Intervention
- Control (No Intervention): The participants randomized to the control arm will receive standard care treatment but will not be exposed to the intervention. In addition to the baseline data collection they will complete online surveys at 6±2 weeks (Post-intervention), 6±1 month, and 12±2 months post study enrollment.

INTERVENTIONS:
Behavioral: mCare PTOA Intervention — The mCare PTOA intervention includes five evidence-based modules that focus on 1) basic joint health following injury, 2) self-management strategies, 3) weight management, 4) physical activity, and 5) occupational management. These educational modules will serve as the primary intervention in this study.
  Arms: Intervention

SUMMARY:
The overall objective of this study is to evaluate the efficacy of the mare telehealth intervention platform and the intervention on patients' readiness to manage osteoarthritis and patient reported outcomes. To accomplish the stated objectives the investigators will conduct a randomized controlled trial. The independent variable will be group (Intervention vs. Control) and the dependent variables will be patient reported knee status (SA1) and readiness to manage arthritis measures (SA2a), as well as activity level (SA2b). We will also compare knowledge about post-traumatic osteoarthritis (PTOA) between groups prior to and following the intervention (SA3).

DETAILED DESCRIPTION:
The Specific Aims of this project are:

Specific Aim 1: Compare the change in patient reported outcomes for knee pain, knee symptoms, and lack of vigorous knee function, from pre-intervention to immediately post-intervention and 6 and 12 months post-intervention, between the intervention group and the control group.

Hypothesis 1: From pre-intervention to post-intervention and 6 and 12 months post-intervention, significant decreases in knee pain, knee symptoms, and lack of vigorous knee function will be observed in the intervention group. However, there will be no significant decreases in these outcomes for control participants.

Specific Aim 2: Compare the proportion of participants that demonstrate changes on intermediate outcomes (increased readiness to manage PTOA and decreased knee loads from discretionary physical activity), from pre-intervention to immediately post-intervention and 6 and 12 months post-intervention, between the intervention group and the control group.

Hypothesis 2a: The proportion of participants that demonstrate an improvement in readiness to manage PTOA risk factors, as indicated by a one-step change on the Readiness to Manage Arthritis Questionnaire, will be significantly higher in the intervention group than in the control group, at 6 and 12 months post-intervention.

Hypothesis 2b: Intervention participants will demonstrate a reduction in recreational activities that place high load on the knee, as indicated by a mean decrease on Marx Activity Scale, that will be significantly larger than any decrease in the control group, immediately post-intervention and at 6- and 12-months post-intervention.

Specific Aim 3: Compare knowledge about osteoarthritis (OA) risk factors between groups pre- and post-intervention.

Hypothesis 3: The proportion of participants that demonstrate knowledge of osteoarthritis pre- and post-intervention will significantly increase in the intervention group compared to the control group post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Current or former United States Military Academy (USMA) cadet or active duty service member who has had at least one Anterior Cruciate Ligament (ACL) surgery

Exclusion Criteria:

* Do not have access to a personal mobile device (tablet or smart phone)
* Are less than 6 months post-surgery
* Known deployment within the next 12 months that would remove them from connectivity with a telehealth application for more than 3 months
* Have not been cleared for full unrestricted return to activity/duty post ACL reconstruction

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Knee Function | pre-intervention, immediately post-intervention (~6-weeks), 6-months Post Intervention, 12 months post intervention
  Knee Injury and Osteoarthritis Outcome Score (KOOS)
Readiness to Manage Arthritis | pre-intervention, immediately post-intervention (~6 weeks), 6 months post-intervention, 12 months post-intervention
  Readiness to Manage Arthritis Questionnaire

SECONDARY OUTCOMES:
Physical Activity | pre-intervention, immediately post-intervention (~ 6-weeks), 6 months post-intervention, 12 months post-intervention
  Marx Activity Rating
OA Knowledge | pre-intervention and immediately post-intervention (~6-weeks)
  OA Knowledge

OTHER OUTCOMES:
Knee Function | pre-intervention, immediately post-intervention (~6-weeks), 6 months post-intervention, 12 months post-intervention
  WOMAC
Measure of Intermittent and Constant Osteoarthritis Pain | pre-intervention, immediately post-intervention (~6-weeks), 6 months post-intervention, 12 months post-intervention
  ICOAP (Intermittent and Constant OA Pain)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Cameron, PhD, Principal Investigator — Keller Army Community Hospital
Locations (1):
- Keller Army Community Hospital, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: No